CLINICAL TRIAL: NCT01958437
Title: Enhancing Spatial Navigation Using Non-Invasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C1381-P
Record Dates: First submitted 2013-09-23; First posted 2013-10-09 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
Keywords: Aging; Alzheimer's Disease/Dementia; Cognitive Disorders; Imaging; Magnetic Resonance Imaging (MRI); Neurology; Physical Medicine & Rehabilitation; transcranial direct current stimulation
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Transcranial Direct Current Stimulation
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Cognitively intact older adults - ACTIVE tDCS (Experimental): Group receives active brain stimulation
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- MCI ACTIVE tDCS (Active Comparator): Group receives active brain stimulation
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Cognitively intact older adults - SHAM tDCS (Sham Comparator): Group receives sham brain stimulation
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- MCI SHAM tDCS (Sham Comparator): Group receives sham brain stimulation
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Active and/or sham; All participants receive both stimulation condition. Groups will be counterbalanced (half receiving active tDCS in the first session and sham in the second session; the other half receiving the opposite).

SUMMARY:
Remembering how to travel from one location to another is critical in everyday life, yet this vital ability declines with normal aging and can be further affected by conditions that disproportionately affect the elderly, such as vision loss or progressive dementia. Human and animal research has shown that two distinct memory systems interact during navigation. The first, referred to as allocentric navigation, is very flexible and uses spatial knowledge of key features or landmarks to develop and use a mental map of the environment. This approach involves brain regions that are critical for new learning and memory but that decline with age. The second, referred to as egocentric navigation, is inflexible and relies on "habit" memories that link specific features with specific directions. This approach relies on brain regions that are critical for "automatic" responses and that are relatively unaffected by age.

The main problem is that allocentric navigation declines with age and is accompanied increased dependence on egocentric navigation. This change increases the risk of becoming disoriented or "lost" when traveling in unfamiliar areas or even when traveling new routes in familiar areas. Therefore, the main goal of this project is to examine whether non-invasive brain stimulation, specifically transcranial direct current stimulation, can improve allocentric navigation in healthy older adults and patients with mild cognitive impairment.

Participants will complete two functional magnetic resonance imaging sessions while learning new environments. Before one of these sessions, participants will receive active brain stimulation over the parietal cortex. Before the other session, participants will receive sham brain stimulation over the parietal cortex. The effects of this stimulation will be evaluated using both an allocentric and an egocentric memory test. Physiologic effects will be evaluated using both task-based and resting-state MRI.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria (all participants):

* All medications stable for approximately 1-2 months;
* No history of severe mental illness;
* No current untreated alcohol or substance abuse/dependence;
* English as native and preferred language;
* MRI-compatible if taking part in fMRI studies
* Able to give informed consent.

MCI Inclusion Criteria:

* Diagnosis of amnestic MCI based on criteria set forth by Petersen (2004). Additionally, other potential causes of cognitive deficit ruled out by the referring physician;

Healthy older adults

* intact cognitive functioning as measured by neuropsychological testing

Exclusion Criteria:

* History of neurological disease or injury
* History of severe mental illness
* Current untreated alcohol or substance abuse
* Other conditions may exclude; please discuss with contact

Ages: 50 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Hampstead, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] England HB, Fyock C, Meredith Gillis M, Hampstead BM. Transcranial direct current stimulation modulates spatial memory in cognitively intact adults. Behav Brain Res. 2015 Apr 15;283:191-5. doi: 10.1016/j.bbr.2015.01.044. Epub 2015 Jan 31. PMID 25647757
- [Derived] Lengu K, Ryan S, Peltier SJ, Tyszkowski T, Kairys A, Giordani B, Hampstead BM. Effects of High Definition-Transcranial Direct Current Stimulation on Local GABA and Glutamate Levels Among Older Adults with and without Mild Cognitive Impairment: An Exploratory Study. J Alzheimers Dis. 2021;84(3):1091-1102. doi: 10.3233/JAD-201091. PMID 34602464

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitively Intact -Active Then Sham tDCS; Cognitively Intact - Sham Then Active; MCI - Active Then Sham; MCI - Sham Then Active: All participants received active and sham transcranial direct current stimulation (tDCS). Participants were randomized to order (i.e., half received active tDCS in the first session and sham in the second session; the other half received the opposite).
Period: Overall Study
Arm/Group | Cognitively Intact -Active Then Sham tDCS | Cognitively Intact - Sham Then Active | MCI - Active Then Sham | MCI - Sham Then Active
Started | 11 | 11 | 11 | 11
Completed | 11 | 11 | 10 | 10
Not Completed | 0 | 0 | 1 | 1
Not completed — Incidental MRI findings | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cognitively Intact Older Adults; Patients With Mild Cognitive Impairment: All participants received active and sham transcranial direct current stimulation (tDCS). Participants were randomized to order (i.e., half received active tDCS in the first session and sham in the second session; the other half received the opposite).
- Total: Total of all reporting groups
Arm/Group | Cognitively Intact Older Adults | Patients With Mild Cognitive Impairment | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.15 (7.14) | 69.5 (6.55) | 70.8 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Accuracy in Centimeters From Target Location for Allocentric
Description: 1 active tDCS; 1 sham tDCS for each measure. Participants touched a screen (using a ELO 19" touchscreen monitor) to document the location of the landmark. The distance between the actual vs. selected location served as the dependent measure.
Time Frame: Outcome assessed after each of 2 sessions (estimated within 1 week of each other)
Population: Computer errors caused missing data for a subset (n=4) of participants; those data have simply been omitted from analyses below.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Groups:
- Cognitively Intact ACTIVE tDCS; MCI ACTIVE tDCS: All participants received active and sham transcranial direct current stimulation (tDCS). Participants were randomized to order (i.e., half received active tDCS in the first session and sham in the second session; the other half received the opposite).
- Cognitively Intact SHAM tDCS; MCI SHAM tDCS: all participants received sham in a randomized order
Arm/Group | Cognitively Intact ACTIVE tDCS | MCI ACTIVE tDCS | Cognitively Intact SHAM tDCS | MCI SHAM tDCS
Number analyzed (Participants) | 22 | 20 | 22 | 20
Centimeters (cm) | 13.24 (3.96) | 15.38 (2.13) | 14.22 (2.78) | 15.03 (1.77)
Statistical Analysis 1: Comparison: Cognitively Intact ACTIVE tDCS vs Cognitively Intact SHAM tDCS; RM ANCOVA (covarying order) for cognitively intact groups; Test type: Superiority; p = .048, ANCOVA
Statistical Analysis 2: Comparison: MCI ACTIVE tDCS vs MCI SHAM tDCS; RM ANCOVA (covarying order) for MCI group; Test type: Superiority; p = .063, ANCOVA

2. Primary Outcome: Hippocampal BOLD Signal During Task-based fMRI
Description: BOLD signal change comparing active to sham tDCS during Allocentric navigation (i.e., active HD-tDCS > sham HD-tDCS). Activation maps thresholded at p<.01 with minimum cluster size of 5 voxels.
Time Frame: change between active and sham tDCS sessions (<1month)
Population: Participants from each group were excluded due to movement artifact that invalidated fMRI data.
Measure: Mean (Standard Deviation); unit: Percent signal change
Groups:
- MCI Sham HD-tDCS; Cognitively Intact ACTIVE HD-tDCS; Cognitively Intact Sham HD-tDCS: All participants received active and sham transcranial direct current stimulation (tDCS). Participants were randomized to order (i.e., half received active tDCS in the first session and sham in the second session; the other half received the opposite).
Arm/Group | MCI ACTIVE tDCS | MCI Sham HD-tDCS | Cognitively Intact ACTIVE HD-tDCS | Cognitively Intact Sham HD-tDCS
Number analyzed (Participants) | 19 | 19 | 19 | 19
Percent signal change | .089 (.12) | .037 (.123) | .143 (.134) | .107 (.117)
Statistical Analysis 1: Comparison: MCI ACTIVE tDCS vs MCI Sham HD-tDCS; Change between active and sham tDCS sessions for allocentric blocks; Test type: Superiority; p = .27, ANCOVA; Main effect of stimulation covarying session order
Statistical Analysis 2: Comparison: Cognitively Intact ACTIVE HD-tDCS vs Cognitively Intact Sham HD-tDCS; Test type: Superiority; p < .001, ANCOVA

3. Primary Outcome: Dorsal Attention Network Connectivity During Resting-state fMRI
Description: Change in resting state functional connectivity strength between active and sham tDCS sessions. Strength is measured by Pearson r correlations between nodes, which are z-transformed, and summated.
Time Frame: change between active and sham tDCS sessions (<1month)
Population: Participants from each group were excluded due to movement artifact that invalidated fMRI data.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- MCI ACTIVE HD-tDCS; Cognitively Intact SHAM HD-tDCS; MCI SHAM HD-tDCS: All participants received active and sham transcranial direct current stimulation (tDCS). Participants were randomized to order (i.e., half received active tDCS in the first session and sham in the second session; the other half received the opposite).
Arm/Group | Cognitively Intact ACTIVE tDCS | MCI ACTIVE HD-tDCS | Cognitively Intact SHAM HD-tDCS | MCI SHAM HD-tDCS
Number analyzed (Participants) | 20 | 18 | 20 | 18
arbitrary units | 29.41 (7.09) | 30.93 (11.97) | 30.39 (8.2) | 31.47 (9.89)
Statistical Analysis 1: Comparison: Cognitively Intact ACTIVE tDCS vs Cognitively Intact SHAM HD-tDCS; Test type: Superiority; p < .001, ANCOVA; Main effect of session using repeated measures ANCOVA covarying stimulation order
Statistical Analysis 2: Comparison: MCI ACTIVE HD-tDCS vs MCI SHAM HD-tDCS; Test type: Superiority; p = .046, ANCOVA; Main effect of session using repeated measures ANCOVA covarying stimulation order

4. Primary Outcome: Egocentric
Description: Number of turns correctly recalled for each egocentric environment
Time Frame: Outcome assessed after each of the 2 sessions
Population: Participants from each group were excluded due to movement artifact that invalidated fMRI data.
Measure: Mean (Standard Deviation); unit: Correct turns
Arm/Group | Cognitively Intact ACTIVE tDCS | MCI ACTIVE tDCS | Cognitively Intact SHAM tDCS | MCI SHAM tDCS
Number analyzed (Participants) | 22 | 20 | 22 | 20
Correct turns | 9.05 (3.53) | 8.21 (3.08) | 9.85 (3.6) | 7.47 (2.53)
Statistical Analysis 1: Comparison: Cognitively Intact ACTIVE tDCS vs Cognitively Intact SHAM tDCS; Repeated Measures ANCOVA (covarying stimulation order); Test type: Superiority; p = .497, ANCOVA
Statistical Analysis 2: Comparison: MCI ACTIVE tDCS vs MCI SHAM tDCS; Test type: Superiority; p = .599, ANCOVA

ADVERSE EVENTS:
Time Frame: duration of each participant's study related activities (~2 weeks), with monitoring ending following the second tDCS session
Description: All participants completed a standardized side effect questionnaire after every tDCS session.
Groups:
- Cognitively Intact Active; Cognitively Intact Sham; MCI Active; MCI Sham: All participants received active and sham transcranial direct current stimulation (tDCS). Participants were randomized to order (i.e., half received active tDCS in the first session and sham in the second session; the other half received the opposite).
Arm/Group | Cognitively Intact Active | Cognitively Intact Sham | MCI Active | MCI Sham
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 13/21 | 17/22 | 15/20 | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitively Intact Active (N=21) | Cognitively Intact Sham (N=22) | MCI Active (N=20) | MCI Sham (N=20)
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Headache
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Neck pain
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (5) — Scalp pain
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 13 (13) | 17 (17) | 8 (8) | 9 (9) — Tingling
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8) | 7 (7) | 8 (8) — Itching
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 11 (11) | 9 (9) | 15 (15) | 12 (12) — Burning
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Skin redness
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) — Sleepiness
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1) — Concentration changes
Side effect questionnaire (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — mood changes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT01958437/Prot_SAP_000.pdf